CLINICAL TRIAL: NCT03353545
Title: A Retrospective Chart Review and a Prospective Study of the POmalidomide Plus LoW Dose Dexamethasone Efficacy in Relapsed/ ReFractory Multiple Myeloma Patients Under Real-Life Conditions,
Brief Title: Retrospective and Prospective Study of POmalidomide Plus LoW Dose Dexa Efficacy in RRMM Patients Under Real-Life Conditions
Acronym: POWERFUL
Status: Completed | Type: Observational
Sponsor: Genesis Pharma S.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-GEN-POM-001
Record Dates: First submitted 2017-10-31; First posted 2017-11-27 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Relapse/Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The importance of real-world evidence studies stems from the following considerations. The study population of a specific clinical trial needs to meet strict inclusion and exclusion criteria, which result in a population of participants that is not necessarily representative of the study population of interest treated in routine care. Furthermore, the outcomes of a clinical trial occur under controlled conditions that do not necessarily reflect the routine healthcare practice. This is especially true among patient populations with challenging to treat disease such as in MM, where personalized therapeutic approaches are commonly considered taking into consideration the patients' age and associated comorbidities, among other factors. In addition, observational studies, due to their non-interventional nature, often show increased degree of heterogeneity across the enrolled patient populations compared to clinical studies, thus aiding generalizability of the results.

In light of the above and due to the scarcity of evidence regarding the outcomes for patients with RRMM receiving Pom/LoDex in routine clinical practice, this retrospective chart review and prospective observational study aims to assess the PFS and response to treatment as well as to obtain real-world evidence on the utilization patterns and management strategy of Pom/LoDex in routine clinical care settings in Greece.

This is a non-interventional, multicenter, single-country, retrospective chart review and prospective cohort study which will include a representative sample of patients with RRMM who have been initiated on Pom/LoDex between 01 January 2016 and 28 February 2019 in the third line and beyond treatment setting under routine care conditions in Greece.

The study will be carried out by hospital-based hematology specialists practicing in geographically diverse locations throughout Greece and will be conducted under real-world conditions of daily clinical practice.

ELIGIBILITY:
* Patients eligible for inclusion in this study have to meet all of the following criteria:

  * Adult subjects (aged ≥18 years) of either gender.
  * Subjects with a documented RRMM diagnosis according to IMWG or EBMT criteria prior to Pom/LoDex treatment.
  * Subjects who have been initiated on Pom/LoDex treatment as per the product's Summary of Product Characteristics (SmPC) between 01 January 2016 and 28 February 2019, after having received at least two prior therapies including both lenalidomide and bortezomib and whose disease progressed after the last treatment.*
  * Note: Retrospective patients who at the time of their enrollment in the study have already completed 3 or more cycles with Pom/LoDex must have available at least one post-baseline response assessment
  * Subjects with available medical files/records and detailed historical data on their disease course and clinical management.
  * Provision of signed informed consent form (ICF) for collecting and analyzing medical data pertinent to the objectives of this study.**

    * Note: For retrospective subjects who are deceased at the date of enrollment into the study a waiver of consent will be requested by the Hospital Scientific Committee and/or Administrative Board of each participating site to either implement a hospital ICF already in place or provide written approval of this study- specific waiver. In the occasion that waiver of consent is not granted by the Scientific Committee and/or Administrative Board of the study site, deceased subjects will not be enrolled in the study.

Exclusion Criteria:

A patient who meets any of the following criteria will be excluded from participation in this study:

* Prior malignancy (within the 3 years preceding initial diagnosis of MM).
* Concurrent administration of anti-cancer regimens for malignancies other than MM.
* Subjects currently participating or who have participated, during the treatment phase, in any investigational program with interventions outside of routine clinical practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 100 adult patients with RRMM who have been initiated on Pom/LoDex treatment as indicated in the product's Summary of Product Characteristics (SmPC) (i.e., after having received at least two prior therapies including both lenalidomide and bortezomib and whose disease progressed after the last treatment) between 01 January 2016 and 28 February 2019 and who are eligible for participation in the study according to the inclusion and exclusion criteria -as outlined in Section 10- are planned to be recruited in the present clinical study. For the justification of the sample size please refer to Section 13.1.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Pom/LoDex in terms of median PFS | median time from start of Pom/LoDex treatment to disease progression or death, through study completion and maximum 50 months
  To evaluate the effectiveness of Pom/LoDex in terms of median PFS, in eligible patients with RRMM in a real world setting in Greece.

SECONDARY OUTCOMES:
Response to Pom/LoDex treatment in terms of ORR | from start of Pom/LoDex until achievement of PR or better, through study completion and maximum 50 months
  To estimate the response to Pom/LoDex treatment in terms of ORR in the study RRMM population
Response to Pom/LoDex treatment in terms of CBR | from start of Pom/LoDex until achievement of MR or better, through study completion and maximum 50 months
  To estimate the response to Pom/LoDex treatment in terms of clinical benefit rate (CBR) in the study RRMM population
Response to Pom/LoDex treatment in terms of DCR | from start of Pom/LoDex until achievement of SD or better, through study completion and maximum 50 months
  To estimate the response to Pom/LoDex treatment in terms of disease control rate (DCR) in the study RRMM population
TTR among the RRMM study population who achieved at least partial response (PR) | median from start of Pom/LoDex to first documented response (TTR), through study completion and maximum 50 months
  To estimate time to response (TTR) to Pom/LoDex among the RRMM study population who achieved at least partial response (PR);
DoR among the RRMM study population who achieved at least partial response (PR) | median from start of Pom/LoDex to first disease progrestion or death (DoR), through study completion and maximum 50 months
  To estimate duration of response (DoR) to Pom/LoDex among the RRMM study population who achieved at least partial response (PR);
12-month PFS rate | time from start of Pom/LoDex until 12 months
  To evaluate the 12-month PFS rate under treatment with Pom/LoDex in the RRMM study population
Time to progression | median time from start of Pom/LoDex until disease progression or death, through study completion and maximum 50 months
  To estimate time to progression (TTP) under treatment with Pom/LoDex in the RRMM study population
Real-world utilization patterns of Pom/LoDex in the RRMM study population | no time frame - only proportion of patients in 12 month follow-up
  To capture the real-world utilization patterns of Pom/LoDex in the RRMM study population, in terms of the rate of its incorporation in the third versus a later-line therapeutic strategy, and the prior treatment modalities employed in real-life clinical practice

OTHER OUTCOMES:
Evaluate the effectiveness and response to Pom/LoDex treatment in the subpopulations of RRMM patients who have been initiated on Pom/LoDex in the third line versus later line setting | from start of Pom/LoDex until 12 month follow-up
  Separation of Pom/Dex treatment outcomes in two subgroups of patients (treated in the third line versus later lines)
To evaluate the improvement of the QoR with Pom/LoDex continued treatment | from start of Pom/LoDex until 12 month follow-up
  To measure the improvement of the quality of response with Pom/LoDex continued treatment over time (i.e. improvement from PR to VGPR)

CONTACTS AND LOCATIONS:
Overall Officials: Kiki Karvounis, Study Director — Genesis Pharma S.A.
Locations (1):
- Ag.Andreas General Hospital, Pátrai, Greece

REFERENCES:
- [Result] Terpos E, Repousis P, Lalayanni C, Hatjiharissi E, Assimakopoulou T, Vassilopoulos G, Pouli A, Spanoudakis E, Michalis E, Pangalis G, Ntanasis-Stathopoulos I, Poziopoulos C, Kyrtsonis MC, Pappa V, Symeonidis A, Georgopoulos C, Zikos PM, Gavriatopoulou M, Papadaki HA, Dadakaridou M, Karvounis-Marolachakis K, Katodritou E. Pomalidomide Plus Low-Dose Dexamethasone in Relapsed/Refractory Multiple Myeloma Patients: Results of the Real-World "POWERFUL" Study. J Clin Med. 2021 Apr 5;10(7):1509. doi: 10.3390/jcm10071509. PMID 33916376